CLINICAL TRIAL: NCT04233047
Title: Fostemsavir Compassionate Use Named Patient Program for the Treatment of Human Immunodeficiency Virus 1 (HIV-1)
Status: Available | Type: Expanded Access
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 207214
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: HIV Infections
Keywords: Human Immunodeficiency Virus 1 (HIV-1)
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — fostemsavir

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Fostemsavir — Fostemsavir 600 mg extended release tablets, administered 600 mg twice daily, will be supplied for compassionate use for the identified individual patient.

SUMMARY:
Compassionate use access to fostemsavir (GSK3684934, formerly BMS-663068) for the treatment of HIV infection in individuals with multidrug resistant HIV-1 infection who are experiencing virologic failure and are unable to comprise a suppressive regimen with currently available antiretrovirals.

Direct inquires to the ViiV Compassionate Use Portal via https://viiv-cu-portal.idea-point.com/

DETAILED DESCRIPTION:
Fostemsavir (FTR) is the prodrug of temsavir (TMR), which is a novel, first-in-class attachment inhibitor being developed as a potential treatment of HIV-1 infection. Investigational FTR is being made available on a compassionate use named patient basis for the treatment of HIV infection in individuals with multidrug resistant HIV-1 infection who are experiencing virologic failure (confirmed HIV-1 RNA ≥1000 c/mL) and are unable to comprise a suppressive regimen with currently available antiretrovirals. Such patients, who are often heavily treatment experienced (HTE), represent a small and highly vulnerable subgroup within the overall HIV patient population. The care of HTE patients is difficult and often complicated by the presence of complex comorbidities, extensive concomitant medication profiles, and advanced HIV disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has given consent for treatment
2. Patient is male or non-pregnant female, age 18 years and older. NOTE: there may be allowance for a lower minimum age if dictated by local regulatory and/or legal requirements.
3. Patient has chronic HIV-1 infection and is heavily treatment experienced
4. Patient is experiencing virologic failure (confirmed HIV-1 RNA ≥1000 c/mL) on a current antiretroviral therapy (ART) regimen and:

   1. is unable to comprise a suppressive regimen without fostemsavir due to documented multi-drug resistance test results and/or intolerance and/or contraindication AND
   2. has no more than 2 fully active ART agents (0, 1, or 2 ART agents) which can be paired with fostemsavir as part of a viable combination ART regimen
5. Patient meets the following reproductive status criteria:

   1. Women must not be breastfeeding
   2. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 24 hours prior to the start of fostemsavir and must agree to periodic pregnancy testing (as per local standard of care) for the duration of treatment with fostemsavir.
   3. WOCBP must agree to use at least 1 method of effective contraception for the duration of treatment with fostemsavir and 60 hours after fostemsavir drug exposure. Males must inform their female partners who are WOCBP of the contraceptive requirements of the NPP to which they too are expected to adhere.
   4. Males who are sexually active with WOCBP must use condoms for the duration of treatment with fostemsavir and 60 hours after last dose. In addition, males must be willing to refrain from sperm donation during this time.
   5. WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements but must comply with the pregnancy testing schedule as outlined in inclusion criterion 5b.

Physicians shall counsel WOCBP and males who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy. At a minimum, contraceptive counselling should be provided at the time of consent.

Exclusion Criteria:

Patients will not be eligible for fostemsavir compassionate use if any of the following criteria apply:

1. Patient is eligible to access commercial fostemsavir or investigational fostemsavir by means other than the named patient program.
2. Patient is taking one or more prohibited medications including:

   1. strong CYP3A inducers including, but not limited to: carbamazepine, phenytoin (anticonvulsants), mitotane (antineoplastic), enzalutamide (androgen receptor inhibitor), rifampicin (antimycobacterial) and St John's wort (Hypericum perforatum, herbal supplement),
   2. elbasvir/grazoprevir (hepatitis C direct acting antiviral)
3. Patient has a prior history of poor adherence with multiple failed attempts of oral ART

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare